CLINICAL TRIAL: NCT03595904
Title: Internet-Based Motivational Interviewing for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sarah Miller, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCO 14-0275; K07CA190726 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal neoplasms; colonoscopy; African Americans; Telemedicine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups (1:1).
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the participants' assigned study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Motivate group (Experimental): Participants complete a 20-minute tablet app, called e-Motivate, and receive usual care.
  Interventions: Behavioral: E-Motivate group
- Usual Care Group (Active Comparator): Participants in the usual care group will receive standard clinical care for patients referred for a screening colonoscopy
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: E-Motivate group — Participants in the e-Motivate group will receive standard clinical care which includes patient navigation (e.g., scheduling and reminders). They will also complete a 20-minute, motivational interviewing informed tablet app in the clinic immediately after they receive a referral for a screening colonoscopy. The tablet app consists of educational videos, interactive exercises (e.g., decisional balance), and personalized feedback (e.g., print summary).
  Arms: E-Motivate group
Behavioral: Usual Care Group — Participants in the usual care group will receive standard clinical care for patients referred for a screening colonoscopy. In particular, they will receive patient navigation which includes scheduling the colonoscopy appointment, making reminder calls, and providing print materials regarding the bowel prep instructions.
  Arms: Usual Care Group

SUMMARY:
Compared to other racial groups, African Americans have the highest colorectal cancer (CRC) morbidity and mortality rates. Although colonoscopies can prevent CRC, nearly one third of African Americans have not received a screening colonoscopy within the recommended time frame (one colonoscopy per ten years). It is critical to increase African Americans' screening colonoscopy rates in order to reduce racial inequities in CRC morbidity and mortality. Previous research suggests that a motivational interviewing based intervention may help improve screening colonoscopy uptake. This study will conduct a randomized clinical trial examining the efficacy of a motivational interviewing informed tablet app, called e-Motivate, to improve African Americans' screening colonoscopy uptake. Participants will be African Americans who receive a referral for a screening colonoscopy. Participants (N=200) will be randomly assigned to one of two groups: (1) usual care group (N=100); or (2) e-Motivate app group (N=100). Participants in the usual care group will receive standard clinical care which includes patient navigation (e.g., scheduling, reminder calls). Participants in the e-Motivate group will complete the e-Motivate app in the clinic immediately after they receive a referral for the screening colonoscopy. The participants in the e-Motivate app group will also receive usual care. Six months following the initial referral, participants' medical charts will be reviewed to determine whether the participants completed the recommended screening colonoscopy. Secondary outcomes (e.g., bowel prep quality, number of cancellations) will also be analyzed.

DETAILED DESCRIPTION:
Colorectal cancer (CRC), a largely preventable disease, remains the third leading cause of cancer death in the United States. Compared to other racial groups, African Americans have the highest CRC morbidity and mortality rates. Recent reports have found that African Americans' CRC incidence rates are 20% higher and mortality rates are 45% higher than those of whites. Given these disparities, it is critical to increase African Americans' participation in CRC screenings. Of the recommended CRC screening mechanisms, a colonoscopy is often the preferred method because it allows for both the detection and removal of precancerous and cancerous polyps. Although screening colonoscopies can detect and prevent CRC, more than 1/3 of African Americans have not received a screening colonoscopy within the recommended time frame (one screening colonoscopy per ten years). It is critical to increase African Americans' screening colonoscopy rates in order to reduce racial inequities in CRC morbidity and mortality.

A motivational interviewing (MI) intervention can help improve African Americans' screening colonoscopy uptake. MI is a brief patient-centered intervention that increases perceived competence, autonomy, and relatedness in order to promote behavioral change. Extensive research supports the efficacy of MI to promote preventive health screening uptake, including increasing screening colonoscopy rates, and MI has proven efficacious with African Americans across a wide range of diseases.

Traditionally, MI is delivered live, where individuals meet with a professional for a one-on-one intervention. Although efficacious, live-MI is not without limitations. Of greatest concern, live-MI requires both staffing and economic resources, limiting its ability to be widely disseminated. A digital intervention, such a tablet app, may overcome these limitations. By eliminating the need for an on-site professional, a tablet app is a high reach, low cost intervention with the potential to have a significant public health impact.

The primary goal of this study is to conduct a randomized clinical trial (RCT) that examines the efficacy of a tablet app, called e-Motivate, to improve screening colonoscopy rates in African Americans.

The app first underwent iterative field-testing and subsequent modifications to ensure that the app had high usability and acceptability ratings.

The final version of the app, called e-Motivate, will be tested in a randomized clinical trial. African American patients referred for a screening colonoscopy will be recruited to the RCT. Participants (N=200) will be randomly assigned to a usual care group (N=100) or an e-Motivate group (N=100). Participants in the usual care group will receive standard patient navigation (e.g., scheduling, reminder calls). Participants in the e-Motivate group will receive standard clinical care and will also complete the e-Motivate app. The app will be a 20-minute tablet app that will include motivational interviewing informed exercises and education. The app will be completed in the clinic immediately after a participant receives a referral for a screening colonoscopy. Six months following the initial referral, participants medical charts will be reviewed to determine whether they completed the recommended screening colonoscopy. It is hypothesized that participants in the e-Motivate group will be more likely to complete the recommended screening colonoscopy.

The study will also explore whether the e-Motivate app can improve secondary outcomes (e.g., bowel prep quality, number of cancellations).

Potential mediators, informed by Self Determination Theory, will be evaluated. Potential moderators (e.g., age, education, family history of CRC) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as African American/Black
* received a referral for a screening colonoscopy
* recommended age to begin screening for colorectal cancer (based on current guidelines)
* English speaking

Exclusion Criteria:

* hearing or vision impaired
* participated in the previous iterative field testing

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Miller, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai and Mount Sinai Hospital
Locations (1):
- Icahn School of Medicine at Mount Sinai and Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller SJ, Foran-Tuller K, Ledergerber J, Jandorf L. Motivational interviewing to improve health screening uptake: A systematic review. Patient Educ Couns. 2017 Feb;100(2):190-198. doi: 10.1016/j.pec.2016.08.027. Epub 2016 Aug 26. PMID 27599713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment sites: Primary care and Gastroenterology clinics in the Mount Sinai Health System. Enrollment started in November 2017 through November 2019.
Groups:
- E-Motivate Group: Participants completed a 20-minute tablet app, called e-Motivate and received usual care. In particular, participants in the e-motivate group completed a 20-minute, motivational interviewing informed tablet app in the clinic after they received a physician referral for a screening colonoscopy. The tablet app consisted of educational videos, interactive exercises (e.g., decisional balance), and personalized feedback (e.g., print summary).
- Usual Care Group: Participants in the usual care group received standard clinical care for patients referred for a screening colonoscopy. In particular, they received patient navigation (e.g., assistance scheduling the screening colonoscopy appointment, making reminder calls, and providing print materials regarding the bowel prep instructions).
Period: Overall Study
Arm/Group | E-Motivate Group | Usual Care Group
Started | 39 | 39
Completed | 29 | 34
Not Completed | 10 | 5
Not completed — Protocol Violation | 3 | 1
Not completed — Deemed medically ineligible for direct access colonoscopy | 4 | 3
Not completed — Insurance complications | 1 | 0
Not completed — COVID-19 halt in non-essential appointments during 6 month follow up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Motivate Group | Usual Care Group | Total
Number analyzed (Participants) | 29 | 34 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.55 (7.42) | 59.15 (7.02) | 58.87 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 44
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 32 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 32 | 58
  White | 0 | 0 | 0
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed a Screening Colonoscopy
Description: Six months following the initial referral, medical charts was reviewed to determine whether the participant completed the recommended screening colonoscopy
Time Frame: six months after the initial referral
Measure: Count of Participants; unit: Participants
Arm/Group | E-Motivate Group | Usual Care Group
Number analyzed (Participants) | 29 | 34
Participants | 19 | 19

2. Secondary Outcome: Number of Participants With Adequate Bowel Prep Quality
Description: An adequate prep which is defined as "adequate, excellent or good". An inadequate prep would be defined as "inadequate, poor or fair". Six months following the initial referral, medical charts was reviewed to determine the physician-rated bowel prep quality for participants who completed the screening colonoscopy.
Time Frame: six months after initial referral
Population: Data only available for those participants with bowel prep quality ratings.
Measure: Count of Participants; unit: Participants
Arm/Group | E-Motivate Group | Usual Care Group
Number analyzed (Participants) | 22 | 19
Participants | 12 | 13

3. Secondary Outcome: Number of Participants Who Had Canceled Appointments
Description: Process variable was assessed via medical chart review six months following the initial referral
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | E-Motivate Group | Usual Care Group
Number analyzed (Participants) | 29 | 34
Participants | 5 | 11

4. Secondary Outcome: Number of Patients Who Had Rescheduled Appointments
Description: Process variable was assessed via medical chart review six months following the initial referral
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | E-Motivate Group | Usual Care Group
Number analyzed (Participants) | 29 | 34
Participants | 0 | 6

5. Secondary Outcome: Number of Participants Who Were No-show Appointments
Description: Process variable was assessed via medical chart review six months following the initial referral
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | E-Motivate Group | Usual Care Group
Number analyzed (Participants) | 29 | 34
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | E-Motivate Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/34
Other Adverse Events (participants affected / at risk) | 0/29 | 0/34

LIMITATIONS AND CAVEATS:
There was notable missing data in the "bowel prep quality" outcome. Not all medical records included a bowel prep quality score. The control condition had 15 missing bowel prep quality ratings and the app condition had 7 missing bowel prep quality ratings. Furthermore, there were inconsistencies in the way in which bowel prep quality was reported (e.g., adequate/inadequate vs. poor, fair, good, excellent).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03595904/Prot_SAP_000.pdf